CLINICAL TRIAL: NCT05174182
Title: A Comparison of Two Different Treatment Approaches for Adolescents With Osgood Schlatter: A Randomized Controlled Superiority Trial (The SOGOOD Trial)
Brief Title: A Comparison of Two Different Treatment Approaches for Adolescents With Osgood Schlatter
Acronym: SOGOOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Aalborg University (Other); University College Copenhagen (Other)
Responsible Party: Principal Investigator, Kasper Krommes, Senior Research Coordinator, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-21028912
Record Dates: First submitted 2021-11-30; First posted 2021-12-30 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Osgood-Schlatter Disease; Apophysitis; Osteochondrosis; Tibia; Physeal Injury
Keywords: Adolescents; Sport; Physical activity; Knee; Load management; Strength training; Accelerometer; Ultrasound; Tibial tubercle; Handheld dynamometry; Handheld algometry; Usual Care
MeSH Terms: conditions — Osteochondrosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: The trial is a single-center pragmatic, double-blinded randomized controlled superiority trial, with a two-group parallel arm design and 1:1 group allocation ratio.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants: Participants are blinded to the actual contents of the two interventions before being allocated, and will remain blinded to the contents of the parallel intervention. They are also blinded to the superiority framework.
  Care provider: Therapists delivering an intervention will likewise be blinded to the contents of the parallel intervention, and to the superiority framework.
  Outcomes assessors: Staff collecting objective outcome data are blinded to group allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A novel treatment approach (Experimental): The experimental intervention were first comprised and tested in a large cohort of 10-14-year-old adolescents with a similar condition (patellofemoral pain) and was associated with a successful outcome after 12 weeks.
  Afterwards, the intervention was changed slightly to target adolescents with Osgood Schlatter and then pilot-tested in a cohort of 51 participants. In this cohort, most participants needed more time to progress through exercises and sport, and the investigators have therefore piloted extending the intervention further in the clinic, with more success on these aspects.
  The experimental intervention will contain an active approach with self-management of load and progressive exercise therapy throughout the treatment course, delivered through 4 one-on-one visits lasting approximately 20 minutes (at months 0, 1, 2, 3) with a physiotherapist and an accompanying leaflet with written and illustrated exercise description, and advice and information.
  Interventions: Other: A novel treatment approach
- Usual care (Active Comparator): The investigators have performed a step-wise mixed-methods sub-study to investigate current standard of care in the most common settings in Denmark (Sports Physiotherapists mainly from private primary practice, and Orthopedic Surgeons caring for these patients, invited from all public secondary care orthopedic departments in Denmark). Results were then combined with reports from patients seen in the clinic (n=34) who were questioned in detail on what modalities and advice they had previously received. The results were mostly compatible with the recent international survey of clinicians treating Osgood-Schlatter. With the findings from this process the investigators have developed a patient-aimed leaflet, which will contain vignettes and elaborations of the multimodal approaches included in the standardized usual care package, which will be implemented through four visits (at months 0, 1, 2, 3) with a physiotherapist (mirroring the plan of care of the experimental group).
  Interventions: Other: Usual care

INTERVENTIONS:
Other: A novel treatment approach — A novel treatment approach, as described before.
  Arms: A novel treatment approach
Other: Usual care — Usual care, as described before.
  Arms: Usual care

SUMMARY:
The most common growth-related injury is Osgood Schlatter, which affects up to 1 in 5 physically active adolescents. It can cause long-term pain and potential discontinuation of sports and physical activity, with sequela well into adulthood. No effective conservative treatments have been documented, and clinical practice is characterized by a wealth of conflicting advice and modalities. A novel treatment approach has shown promising results in a small single-cohort study. Therefore, this study aims to compare this novel treatment with usual care in 10-16-year-old adolescents with Osgood Schlatter.

This single-center pragmatic, double-blinded, randomized, controlled superiority trial, will have a two-group parallel arm design. Participants will undergo 3 months of treatment, followed by 2 months of self-management with self-reported knee function (KOOS-child 'Sport/rec') at 5 months as the primary endpoint.

This trial comparing a novel treatment with usual care for adolescents with Osgood Schlatter could result in an evidence-based treatment ready for implementation in clinical practice, benefitting patients outcomes and clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Tenderness on palpation of the tibial tuberosity or pain during resisted isometric knee extensions
* Insidious onset of pain or swelling of the tibial tuberosity for ≥6 weeks
* Provoked by at least 2 of the following positions or activities; prolonged sitting or kneeling, squatting, running, hopping/jumping, stair walking or during multidirectional sports
* Clinical diagnosis of Osgood Schlatter
* Markedly reduced sports participation OR severely affected by pain during sports participation

Exclusion Criteria:

* Other primary pathology or complaints from other structures of the knee
* Other injuries, complaints or illnesses that may cause disability, or specifically restricts levels of physical activity or sports participation
* Previous surgery in the lower extremities or lumbar spine
* Congenital deformities, device implants og cysts og tumors of the knee
* Participants not willing to cease concomitant treatment
* Participants and their parents not able to understand and communicate in written and verbal Danish

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Knee and Osteoarthritis Outcome Score for Children (KOOS-Child) 'Sport / Recreation' subscale change from baseline | 5 months (secondary timepoints: month 1, 2, 3, 8, 10, 12, 24, 48)
  The scale contains 7 questions answered through a 0-4 likert scale. The scale is normalized to a 0-100 score with 100 be, with zero representing extreme knee problems and 100 representing no knee problems.

SECONDARY OUTCOMES:
Patient Acceptable Symptom State change from baseline | 5 months
  The question pertaining to Patient Acceptable Symptom State (PASS) are designed in collaboration with patient representatives. The recall period will be one week, and the outlook period a 'few months' as in previous applications in musculoskeletal conditions with fluctuating symptoms:
  "If you consider your knee pain during the past week, and how it affects your ability to do activities of daily living (for example participating in school, in sports, and socially), would you consider your current symptom state acceptable for the next few months?". The proportions of yes/no in each group will be captured
Knee and Osteoarthritis Outcome Score for Children (KOOS-Child) 'Quality of Life' Subscale change from baseline | 5 months
  The scale contains 6 questions answered through a 0-4 likert scale. The scale is normalized to a 0-100 score with 100 be, with zero representing extreme knee problems and 100 representing no knee problems.
Frequency of Pain Flares | 5 months
  Weekly average of pain flares over a 4-week period leading up to the 5 months visit. Pain flares are defined as episodes of of 4 or more on the 0-10 numerical pain rating scale with 0 being no pain and 10 being worst pain imaginable.
Pain Flare Intensity change from baseline | 5 months
  Pain intensity as defined as the highest rating of pain on the 0-10 numerical pain rating scale with 0 being no pain and 10 being worst pain imaginable.
Hours of Sports Participation | 5 months
  The level of participation in sports will be captured through weekly monitoring. Participants will be asked if they have been participating in sports in the preceding week, and for how many hours. A 4-week average leading up to the 5 month visit will be calculated
Hours of Physical Activity | 5 months
  Minutes of Moderate to Vigorous Physical Activity (MVPA) will be captured using waterproof 3 axis 12 Hz accelerometers (SENS®, Copenhagen, Denmark) applied once to the participants thigh during the enrollment visit using an adhesive patch. A 4-week average leading up to the 5 month visit will be calculated
  According to WHO recommendations a daily minimum of 60 min of MVPA is needed to stay healthy for 5-17 year olds.Thus being at either under or above this cutoff during a 4-week average leading up to the 5 month visit will be assessed, in addition to a continuous comparison between the two groups of minutes of MVPA during the same time period.
Satisfaction with extent of sports participation change from baseline | 5 months
  Participants will also be asked during clinical visits if they are satisfied with the current extent of their sports participation (Yes/No questions).
Tendinosis signs change from baseline | 5 months
  Involvement of the tendon is common in patients with Osgood Schlatter. Signs of tendinosis will be assess through ultrasound scanning by evaluating either the tendon as thickened or with hyperemia through color-doppler mode.
Infrapatellar bursitis signs change from baseline | 5 months
  In Osgood-Schlatter patients, associated signs of bursitis have shown to be prognostic of a worse outcome. Signs of tendinosis will be assess through ultrasound scanning by evaluating either the infrapatellar bursa as thickened or with hyperemia through color-doppler mode.
Flaviis composite severity score change from baseline | 5 months
  In Osgood-Schlatter patients, gradings of severity have shown to be prognostic of a worse outcome. Severity will be graded according to the ad modum Flaviis 1-4 grading, or as 'normal'.
Anterior Knee Pain Provocation test change from baseline | 5 months
  Adolescents will rate their pain from performing the Anterior Knee Pain Provocation test on the 0-10 numerical pain rating scale with 0 being no pain and 10 being worst pain imaginable.
Pain during knee extension strength test change from baseline | 5 months
  Adolescents will rate pain experienced during a maximal isometric knee extension strength test on the 0-10 numerical pain rating scale with 0 being no pain and 10 being worst pain imaginable.
Pressure-pain threshold at the tibial tubercle change from baseline | 5 months
  To evaluate local hyperalgesia specifically at the tibial tubercle, handheld algometry will be used to detect the pressure (kPa) needed to evoke pain (going from no pain to the slightest sensation of pain) on the tibial tubercle on both knees
Maximal isometric knee extension strength change from baseline | 5 months
  To evaluate the capacity of the quadriceps femoris muscle inserting at the site of pain, handheld dynamometry will be used to measure maximal isometric force generation which will be normalized to bodyweight and lever-length (Nm/kg).
Countermovement jump height change from baseline | 5 months
  As a measure of sports-specific skill, a countermovement jump will be performed to record jump height (cm), using high-speed video analysis via a smartphone app (My Jump 2).
Global rating of Change | 5 months
  To assess patient-assessed improvement or worsening, study personnel will ask participants to rate their perceived level of change from their first visit on a 7-point likert scale ranging from 'Much worse' to 'Much better'.
Patient-specific function scale change from baseline | 5 months
  Study personnel will ask participants to rate their problems with an important activity using the Patient-Specific Functional Scale. They are asked to name a single important activity of their own choosing. Participants then rate their functional limitation with activity on a 0 to 10 scale, where 0 corresponds to being unable to perform activity and 10 is being able to perform activity at same level as before knee pain.
Kinesiophobia change from baseline | 5 months
  To capture level of kinesiophobia, that is, the fear of pain due to movement or exercise, a type of fear-avoidance behavior, the patient-reported 17-item Tampa Scala of Kinesiophobia (TSK-17) will be used.
Self-rated health change from baseline | 5 months
  Self-rated health will be collected through the 0-100 VAS for general health.

OTHER OUTCOMES:
Knee and Osteoarthritis Outcome Score for Children (KOOS-Child) 'Pain' Subscale change from baseline | 5 months
  The scale contains 8 questions answered through a 0-4 likert scale. The scale is normalized to a 0-100 score with 100 be, with zero representing extreme knee problems and 100 representing no knee problems.
Level of pain/discomfort change from baseline | 5 months
  Using the EQ-D5-Y scale, participants are asked on a 3-point likert scale ranging from 1 (I have no pain or discomfort), to 3 (I have extreme pain or discomfort).
Level of sports participation compared to before knee pain | 5 months
  Participants are asked if they perform either 1) at a higher level than before onset of knee pain, 2) at the same level as before onset of knee pain, or 3) at a lower level than before onset of knee pain
Level of physical activity compared to before knee pain | 5 months
  Participants are asked if they are either 1) more physically active than before onset of knee pain, 2) just as physically active as before onset of knee pain, or 3) are less physically active as before onset of knee pain
Time to return to sport | 5 months
  For the subgroup of participants not being active in sports at baseline, the week in which they return to sports participation will be recorded and compared between groups.
Hyperemia of the tibial tubercle change from baseline | 5 months
  Hyperemia of the tibial tubercle will be assess through ultrasound scanning by evaluating hyperemia ad modum Öhberg 1-4 through color-doppler mode.
Palpation pain of the tibial tubecle | 5 months
  Known pain when palpating the tibial tubecle during clinical examination change from baseline
Pain during Countermovement Jump Test change from baseline | 5 months
  Adolescents will rate pain experienced during the CMJ test on the NPRS 0-10.
Countermovement jump power change from baseline | 5 months
  As a measure of power, a countermovement jump will be performed to record jump and power-production (watts), using high-speed video analysis via a smartphone app (My Jump 2).
Knee extensor flexibility change from baseline | 5 months
  Between-group change in knee flexion angle, assessed by smartphone-inclinometry during a modified Thomas Test will be compared.
Satisfaction with treatment | 5 months
  Participants are asked if they believe the treatment recieved have been succesful or not (Yes/No question)
Problems with usual activities change from baseline | 5 months
  Using the EQ-D5-Y scale, participants are asked on a 3-point likert scale ranging from 1 (I have no problems performing my usual activities), to 3 (I am unable to perform my usual activities).
Knee and Osteoarthritis Outcome Score for Children (KOOS-Child) 'Symptoms' change from baseline | 5 months
  The scale contains 7 questions answered through a 0-4 likert scale. The scale is normalized to a 0-100 score with 100 be, with zero representing extreme knee problems and 100 representing no knee problems.
Harms and adverse events | 5 months
  Potential harms and adverse events will be assesed through open-ended questioning during clinical visits in order to assess if further examination or treatment is warranted, and to classify events according to the severity on from Grade 1-5 Using the Common Terminology Criteria for Adverse Events (CTCAE) grading:
  1. Mild: Asymptomatic or minor symptoms; clinical or diagnostic observations only; no intervention needed
  2. Moderate: Minimal, local, or non-invasive intervention indicated
  3. Severe: Medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling
  4. Life-threatening consequences (i.e., immediate risk of death); urgent intervention indicated
  5. Death related to adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Kasper Krommes, Study Director — Amager Hospital
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
To increase transparency and dissemination, all statistical code and fully anonymized dataset will be shared to a open-access repository (such as YODA, Zenodo or Figshare) with a digital objective identifier once all planned publications are accepted or published as pre-print.
  Publication-specific datasets will potentially be posted along with published manuscripts in line with journal policies. If full anonymity cannot be achieved by removing unique data and identifies, a synthetic dataset will be created which will mimic the original dataset by preserving the statistical properties and the relationships between variables.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: All statistical code and fully anonymized dataset will be shared to a open-access repository (such as YODA, Zenodo or Figshare) with a digital objective identifier once all planned publications are accepted or published as pre-print. Anticipated to be before december 1st 2025.
Access Criteria: No criteria, as data will be open access once published.

REFERENCES:
- [Derived] Krommes K, Thorborg K, Clausen MB, Rathleff MS, Olesen JL, Kallemose T, Holmich P. Self-management including exercise, education and activity modification compared to usual care for adolescents with Osgood-Schlatter (the SOGOOD trial): protocol of a randomized controlled superiority trial. BMC Sports Sci Med Rehabil. 2024 Apr 20;16(1):89. doi: 10.1186/s13102-024-00870-0. PMID 38643184

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT05174182/Prot_SAP_001.pdf